CLINICAL TRIAL: NCT06775210
Title: The Effect of Implementing Sleep Care Bundle on Critical Care Nurses' Practice and Patients' Outcomes
Brief Title: Effect of Implementing Sleep Care Bundle on Nurses' Practice and Patients' Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayat Mohamed Fahmy Mohamed Elsheikha, Assistant Lecturer, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sleep Care Bundle
Record Dates: First submitted 2025-01-04; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Ilness; Respiratory Distress Syndrome, Adult
Keywords: sleep care bundle; nursing practice; patients outcomes
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Patient Care Bundles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bundle group (Experimental): receive sleep bundle at sleep
  Interventions: Other: care bundle
- Control group (Placebo Comparator): receive routine care
  Interventions: Other: supportive sleep care

INTERVENTIONS:
Other: supportive sleep care — sleep bundle
  Arms: Control group
Other: care bundle — sleep bundle
  Arms: bundle group

SUMMARY:
Sleep is a fundamental physiological requirement for the human body to heal and overcome an illness or injury . Good sleep is essential for patient recovery and restoration of normal daily functions . Critically ill patients often experience poor sleep quality due to shortened sleep times, increased daytime sleep, and disrupted circadian rhythm . Poor sleep quality is one of the most common complaints of patients who survive their critical illness. Patients' complaints include trouble initiating and maintaining sleep and frequent awakenings with difficulty returning to sleep

DETAILED DESCRIPTION:
Sleep plays an important role in restoring the health of individuals who are ill or injured and essential for critical illness recovery. Poor sleep quality during hospitalization may lead to post-hospital symptoms and increase readmission rates and mortality . Sleep disruption is associated with immune system dysfunction, decreased resistance to infection, changes in nitrogen balance, and impaired wound healing. Therefore, using a standardized non-pharmacological sleep promotion strategy as a sleep care bundle is proposed to reduce the incidence of delirium and improve sleep quality. Internationally, investigations performed to evaluate the effect of implementing sleep care bundle on patients' outcomes had reported its effectiveness. However, studies that addressed the effectiveness of implementing sleep care bundle on critical care nurses' practice and patients' outcomes in Egypt are scarce. Moreover, from our empirical observations, investigators found that there are no available standards of sleep care in the study setting. Furthermore, most nurses do not realize the importance of good sleep for critically ill patients. Therefore, the present study will be carried out to address this issue. Hopefully, the current investigation might generate attention and motivation for using this bundle and for conducting further research studies in this area.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria

* Adult patients of ≥ 18 years old.
* Fully consciousness (Glasgow coma scale score 15; orientation to person, place, and time).
* Spent at least 3 full nights in the above-mentioned ICUs.

Exclusion Criteria:

History of sleep disorder as insomnia and sleep apnea.

* History of mental disorders.
* Patients who are on sedative or narcotic drugs.
* Patients who have visual or hearing impairment.
* History of skin diseases (e.g., contagious skin, eczema).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Sleep Quality Assessment Scale | from first day on admission to three days
  This part used to measure patients' sleep quality. This instrument was developed and validated for ICU patients. It measures participants' perceptions of their sleep in five dimensions: sleep depth, sleep latency (time to fall a sleep), number of awakenings, efficiency (percentage of time awake), and sleep quality. Answers are recorded on a visual analogue scale of 100 mm, with higher scores representing better sleep
Sleep Care Bundle Observation Checklist | Each participant nurse was interviewed individually to gather the demographic characteristics. Nurses' practices regarding the sleep care bundle were observed .
  This part will be developed by the researcher after revising related literature. It will be used to assess nurses' practice regarding implementing the sleep care bundle which encompasses three main domains including; seeing, sensing, and hearing. The intervention that is done correctly will be scored with 1 point while the item that is done incorrectly or not done will be scored with zero point.
Intensive Care Delirium Screening Checklist (ICDSC) | from first day on admission to three days
  This part was adopted from Bergeron, Dubois, Dumont, Dial, & Skrobik (2001) to assess ICU-acquired delirium. Designed for rapid observations from bedside clinical staff routinely gathered throughout a shift. The ICDSC is composed of 8 items including; altered level of consciousness, inattention, disorientation, hallucination or delusion, psychomotor agitation or retardation, inappropriate mood or speech, sleep/wake cycle disturbance, and symptom fluctuation. Patients scored one point for each symptom exhibited during the study and zero points if the symptom did not present.
  The score is ranked as follows:
  * A 0 score indicates that the patient has no delirium
  * A score from 1-3 indicates sub-syndromal delirium
  * A score from 4-8 indicates delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided